CLINICAL TRIAL: NCT02833532
Title: A Multi-center, Randomized, Subject Blind, Active Controlled Design Clinical Study to Evaluate the Efficacy and Safety of Volus as Compared to PowerFill® for Temporary Penile Enhancement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Collaborators: Associacio catalana per a la recerca oncologica i les seves implicacions sanitaries i socials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-Volus-01
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2016-07

CONDITIONS: Penile Enhancement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volus (Experimental): Maxium: 22ml
  Interventions: Device: Volus/Powerfill
- Powerfill (Active Comparator): Maxium: 22ml
  Interventions: Device: Volus/Powerfill

INTERVENTIONS:
Device: Volus/Powerfill — Maximum: 22ml

SUMMARY:
The purpose of this study is to evaluate non-inferial study of the after using Volus application, compared to the powerfill.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged above 20 and below 65. (20≤male≥65)
2. be rating himself, when screening, as "Small or Very Small" on Self-Questioned Questionnaire ( SQQ) including the question: " How do you rate your penile size? // Very small, Small, Normal, Big, Very Big?"
3. During the study period, subjects will not received any treatments associated with penile enhancement.
4. Subjects will sign an informed consent form

Exclusion Criteria:

1. Prior treatment for penile enhancement (e.g. fat, dermal graft).
2. Subjects who have penile malformation (e.g. Peyronie's disease), which can make impossible to perform the intervention
3. Allergic to hyalluronic acid.
4. Inflammatory or/and infectious disease on penis that can affect on this study

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
the Penile Circumference difference at 24 weeks from Baseline value after using Volus application, compared to the Control. | baseline, 24 weeks
  Penile Circumference: The average of Distal-, Mid-, and Proximal-penis measurements when relaxed by tape measurement. Baseline value: Measured baseline length before the intervention.

SECONDARY OUTCOMES:
The Difference in Penile Circumference (each to be measured) at 4, 12 weeks (post last treatment) from Baseline value after using Volus application, compared to the Control. | baseline, 4 weeks, 12 weeks, 24 weeks
The Difference in 5-point scale of penile appearance (each to be measured) at 4, 12, 24 weeks (post last treatment) from Baseline value after using Volus application, compared to the Control. | baseline, 4 weeks, 12 weeks, 24 weeks
The Difference in 5-point scale of sexual satisfaction (each to be measured) at 12, 24 weeks (post last treatment)from Baseline value after using Volus application, compared to the Control. | baseline, 12 weeks, 24 weeks
The Difference in penile length† (each to be measured) at 4, 12, 24 weeks (post last treatment) from ‡B after using Volus application, compared to the Control. | baseline, 4 weeks, 12 weeks, 24 weeks
  † penile length: A length of penile distribution measured from the ventral side of pubo-penile skin junction to the apex of prepuce when relaxed using a tape( or stick)- measure.

CONTACTS AND LOCATIONS:
Locations (1):
- HUGEL, Seoul, South Korea

REFERENCES:
- [Derived] Yang DY, Ko K, Lee SH, Lee WK. A Comparison of the Efficacy and Safety Between Hyaluronic Acid and Polylactic Acid Filler Injection in Penile Augmentation: A Multicenter, Patient/Evaluator-Blinded, Randomized Trial. J Sex Med. 2019 Apr;16(4):577-585. doi: 10.1016/j.jsxm.2019.01.310. Epub 2019 Mar 2. PMID 30833149